CLINICAL TRIAL: NCT02521025
Title: The Impact of Continuous Versus Intermittent Feeding on Changes in Insulin Sensitivity During Bed-rest
Brief Title: Bedrest, Feeding Pattern, and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC 15-3-035
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Atrophy, Disuse; Insulin Resistance
MeSH Terms: conditions — Muscular Disorders, Atrophic; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent feeding (Experimental): Intermittent feeding pattern throughout the bedrest period, with 4 boluses per day
  Interventions: Other: Intermittent feeding pattern
- Continuous feeding (Experimental): Continuous feeding pattern throughout the bedrest period, with 4 boluses per day, without breaks in food supply.
  Interventions: Other: Continuous feeding pattern

INTERVENTIONS:
Other: Intermittent feeding pattern — Intermittent feeding
  Arms: Intermittent feeding
Other: Continuous feeding pattern — Continuous feeding
  Arms: Continuous feeding

SUMMARY:
In the present study, the investigators will assess the impact of two different feeding patterns (continuous vs intermittent) on insulin sensitivity and muscle mass following bedrest.

DETAILED DESCRIPTION:
In the present study, the investigators will assess the impact of two different feeding patterns on insulin sensitivity and muscle mass following bedrest. Healthy, young males will be fed in a continuous (no breaks in food supply) or intermittent (in boluses throughout the day) manner.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 35
* Recreationally active

Exclusion Criteria:

* Type 2 diabetes
* Performing progressive resistance training in 6 months prior to study
* Back/knee/leg problems
* Hypertension
* Use of certain anticoagulants
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs
* Blood donation in past 3 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity (measured as glucose infusion rate during hyperinsulinaemic-euglycaemic clamp) | 7 days bedrest

SECONDARY OUTCOMES:
Change in muscle mass (measured as upper leg muscle cross-sectional area with CT scan) | 7 days bedrest
  Via single-slice CT scan
Change in lean tissue (measured via DEXA scan) | 7 days bedrest
  Via DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Principal Investigator — Maastricht University Medical Centre+
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gonzalez JT, Dirks ML, Holwerda AM, Kouw IWK, van Loon LJC. Intermittent versus continuous enteral nutrition attenuates increases in insulin and leptin during short-term bed rest. Eur J Appl Physiol. 2020 Sep;120(9):2083-2094. doi: 10.1007/s00421-020-04431-4. Epub 2020 Jul 10. PMID 32651634
- [Derived] Dirks ML, Miotto PM, Goossens GH, Senden JM, Petrick HL, van Kranenburg J, van Loon LJC, Holloway GP. Short-term bed rest-induced insulin resistance cannot be explained by increased mitochondrial H2 O2 emission. J Physiol. 2020 Jan;598(1):123-137. doi: 10.1113/JP278920. Epub 2019 Dec 26. PMID 31721213
- [Derived] Dirks ML, Smeets JSJ, Holwerda AM, Kouw IWK, Marzuca-Nassr GN, Gijsen AP, Holloway GP, Verdijk LB, van Loon LJC. Dietary feeding pattern does not modulate the loss of muscle mass or the decline in metabolic health during short-term bed rest. Am J Physiol Endocrinol Metab. 2019 Mar 1;316(3):E536-E545. doi: 10.1152/ajpendo.00378.2018. Epub 2019 Jan 15. PMID 30645176